CLINICAL TRIAL: NCT06830070
Title: Subjective Pain Scoring for Subtenonal Anesthesia During Vitrectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of department, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: SPS
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Epiretinal Membranes; Retinal Detachment; Full Thickness Macular Hole
Keywords: subjective pain score; VAS; subtenonal anesthesia
MeSH Terms: conditions — Epiretinal Membrane; Retinal Detachment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vitreoretinal surface diseases: patients with the indications epiretinal membranes or full thickness macular holes are belonging to the Group of vitreoretnal surface diseases
  Interventions: Other: subjective pain score assessment
- retinal detachment: patients with the indication retinal detachment are belonging to this group
  Interventions: Other: subjective pain score assessment

INTERVENTIONS:
Other: subjective pain score assessment — a questionnaire assessing subjective pain during surgery, using the Visual Analogue Scale with values from 0 to 10

SUMMARY:
Subtenonal anesthesia is a well-known technique of local anesthesia for patients undergoing pars plana vitrectomies. It was described to be efficient with respect to anesthesia of the eye and it showed less risks compared to retrobulbar or parabulbar anesthesia. Purpose of the study is to assess subjective pain scores of patients, that underwent vitrectomy with subtenonal anesthesia.

DETAILED DESCRIPTION:
Subtenonal anesthesia is a well-known technique of local anesthesia for patients undergoing pars plana vitrectomies. It was described to be efficient with respect to anesthesia of the eye and it showed less risks compared to retrobulbar or parabulbar anesthesia. Subjective pain scores of patients, that underwent vitrectomy with subtenonal anesthesia, are probably different among patients with excessive indentation of the bulbus for retinal detachment repair, compared to patients undergoing vitrectomy with membrane peeling for epiretinal membranes or full thickness macular holes. Purpose of the study is to assess subjective pain scores of patients, that underwent vitrectomy with subtenonal anesthesia.

ELIGIBILITY:
Inclusion criteria

* Vitrectomy with subtenonal anesthesia in the time-period from 1.12.2022 to 31.8.2023
* Indication for surgery: retinal detachment, epiretinal membrane, or full thickness macular hole
* Questionnaire for subtenonal anesthesia was already answered by the patients
* Age 18 and older

Exclusion criteria

Any of the following will exclude a subject from the study:

* Surgery in general anesthesia
* Questionnaire missing or incomplete

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having undergone vitrectomy in subtenon´s anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
subjective pain score during surgery | assessed within 24 hours sfter surgery
  subjective pain score during surgery are assessed with Visual Analogue Scale from 0 to 10. The value of 0 represents no pain and the value of 10 represents the highest pain that can be imagined.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Study Chair — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Hindy N, Johnston RL, Jaycock P, Eke T, Braga AJ, Tole DM, Galloway P, Sparrow JM; UK EPR user group. The Cataract National Dataset Electronic Multi-centre Audit of 55,567 operations: anaesthetic techniques and complications. Eye (Lond). 2009 Jan;23(1):50-5. doi: 10.1038/sj.eye.6703031. Epub 2008 Mar 14. PMID 18344970
- [Background] Lai MM, Lai JC, Lee WH, Huang JJ, Patel S, Ying HS, Melia M, Haller JA, Handa JT. Comparison of retrobulbar and sub-Tenon's capsule injection of local anesthetic in vitreoretinal surgery. Ophthalmology. 2005 Apr;112(4):574-9. doi: 10.1016/j.ophtha.2004.10.043. PMID 15808246
- [Background] Friedberg MA, Spellman FA, Pilkerton AR, Perraut LE Jr, Stephens RF. An alternative technique of local anesthesia for vitreoretinal surgery. Arch Ophthalmol. 1991 Nov;109(11):1615-6. doi: 10.1001/archopht.1991.01080110153055. PMID 1845110